CLINICAL TRIAL: NCT00717093
Title: A Randomized, Multicenter, Double Blind, Placebo Controlled Study Evaluating The Efficacy Of Varenicline In Cessation Of Oral Smokeless Tobacco Use
Brief Title: Study Evaluating The Efficacy Of Varenicline In Cessation Of Oral Smokeless Tobacco Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051104
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2010-05-18 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Varenicline Tartrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline Tartrate — Subjects will be up-titrated during the first week of treatment in the following manner: 0.5 mg once daily for 3 days followed by 0.5 mg twice daily for 4 days, and then 1 mg twice daily for the following 11 weeks of the treatment period.
  Other Names: Champix, Chantix, CP-526,555
  Arms: Active
Drug: Placebo — Subjects will be up-titrated during the first week of treatment in the following manner: 0.5 mg once daily for 3 days followed by 0.5 mg twice daily for 4 days, and then 1 mg twice daily for the following 11 weeks of the treatment period.
  Arms: Placebo

SUMMARY:
The primary goal of this study is to compare efficacy of varenicline to placebo for cessation of use of smokeless tobacco.

ELIGIBILITY:
Inclusion Criteria:

* Male or female daily smokeless tobacco users aged 18 years and older, who are motivated to stop use of all tobacco products.
* Subjects must be daily users of nicotine containing smokeless tobacco and using smokeless tobacco on at least 8 occasions per day averaged over a week.
* Have used smokeless tobacco for at least 1 year prior to screening with no period of abstinence >3 months in the past year.

Exclusion Criteria:

* Subjects using nicotine containing products (including smoking tobacco) other than smokeless tobacco for 3 months prior to screening.
* Subjects with exhaled Carbon Monoxide (CO) >10 ppm at baseline.
* Subjects who have used varenicline, bupropion, or NRT within 3 months of screening.
* Subjects currently or within the past 12 months requiring treatment for depression or have a current or prior history of panic disorder, psychosis, bipolar disorder or any other serious mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Norway (7):
  - Pfizer Investigational Site, Florø
  - Pfizer Investigational Site, Hafrsfjord
  - Pfizer Investigational Site, Hamar
  - Pfizer Investigational Site, Hønefoss
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Rådal
  - Pfizer Investigational Site, Trondheim
- Sweden (9):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Jarfalla
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Södertälje
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Sundsvall
  - Pfizer Investigational Site, Umeå

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Fagerstrom K, Gilljam H, Metcalfe M, Tonstad S, Messig M. Stopping smokeless tobacco with varenicline: randomised double blind placebo controlled trial. BMJ. 2010 Dec 6;341:c6549. doi: 10.1136/bmj.c6549. PMID 21134997
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051104&StudyName=Study%20Evaluating%20The%20Efficacy%20Of%20Varenicline%20In%20Cessation%20Of%20Oral%20Smokeless%20Tobacco%20Use

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects will be up-titrated with a matching placebo during the first week of treatment in the following manner: 0.5 mg once daily for 3 days followed by 0.5 mg twice daily for 4 days, and then 1 mg twice daily for the following 11 weeks of the treatment period.
Period: Overall Study
Arm/Group | Varenicline Tartrate | Placebo
Started | 214 | 218
Received Treatment | 213 | 218
Completed | 170 | 170
Not Completed | 44 | 48
Not completed — Adverse Event | 19 | 9
Not completed — Lack of Efficacy | 3 | 13
Not completed — Lost to Follow-up | 9 | 6
Not completed — Withdrawal by Subject | 12 | 19
Not completed — Other | 0 | 1
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline Tartrate | Placebo | Total
Number analyzed (Participants) | 213 | 218 | 431
Age, Customized [Number; unit: participants]
  18 - 44 years | 117 | 115 | 232
  45 - 64 years | 88 | 93 | 181
  >= 65 years | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 189 | 196 | 385

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a 4 Week Continuous Quit Rate (CQR) From Smokeless Tobacco
Description: Number of subjects who reported no use of nicotine-containing products by answering "No" to the nicotine use inventory (NUI) question: Has the subject used any nicotine-containing products in the last 7 days (Week 9) or since last study visit (Week 10 through 12) and confirmed salivary cotinine <= 15 ng/mL.
Time Frame: Weeks 9 through 12
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Varenicline Tartrate | Placebo
Number analyzed (Participants) | 213 | 218
participants | 125 | 85
Statistical Analysis 1: Comparison: Varenicline Tartrate vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-values obtained from logistic regression model including main effects of treatment and center; Missing salivary cotinine values imputed as negative; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.59 to 3.58] — Odds ratio obtained from logistic regression model including main effects of treatment and center

2. Secondary Outcome: Number of Subjects With Continuous Abstinence (CA) of Smokeless Tobacco Use
Description: Number of subjects who remainded abstinent from the period defined as start of the primary endpoint (Week 9) through the end of follow up (Week 26) by reporting no use of nicotine-containing products and confirmed salivary cotinine <= 15 ng/mL.
Time Frame: Week 9 through 12, Week 26
Population: ITT
Measure: Number; unit: participants
Arm/Group | Varenicline Tartrate | Placebo
Number analyzed (Participants) | 213 | 218
participants
  Week 9 | 140 | 101
  Week 10 | 135 | 96
  Week 11 | 132 | 93
  Week 12 | 125 | 85
  Week 26 | 95 | 73
Statistical Analysis 1: Comparison: Varenicline Tartrate vs Placebo; Week 26; Test type: Superiority or Other; p = 0.0118, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and center; Missing salivary cotinine values were imputed as negative; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.12 to 2.58] — Odds Ratio obtained from a logistic regression model including the main effects of treatment and center

3. Secondary Outcome: Number of Subjects With Long Term Quit Rate (LTQR) of Smokeless Tobacco
Description: Number of subjects who were responders for the primary endpoint (4-week CQR for Weeks 9 through 12) and who had no more than 6 cumulative days of using nicotine containing products from Week 12 through Week 26.
Time Frame: Week 26
Population: ITT
Measure: Number; unit: participants
Arm/Group | Varenicline Tartrate | Placebo
Number analyzed (Participants) | 213 | 218
participants | 102 | 78
Statistical Analysis 1: Comparison: Varenicline Tartrate vs Placebo; Test type: Superiority or Other; p = 0.0063, Regression, Logistic; Missing salivary cotinine values were imputed as negative; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.17 to 2.67]

4. Secondary Outcome: Number of Subjects With 7-day Point Prevalence (PP) of Abstinence at the End of Treatment (Week 12) and at the End of Study (Week 26)
Description: Number of subjects at Week 12 and Week 26 reporting no use of nicotine-containing products in the last 7 days and confirmed salivary cotinine <= 15 ng/mL.
Time Frame: Week 12, Week 26
Population: ITT
Measure: Number; unit: participants
Arm/Group | Varenicline Tartrate | Placebo
Number analyzed (Participants) | 213 | 218
participants
  Week 12 | 123 | 85
  Week 26 | 102 | 88
Statistical Analysis 1: Comparison: Varenicline Tartrate vs Placebo; Week 12; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and center; Missing salivary cotinine was imputed as negative; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.52 to 3.41] — Odds ratio obtained from a logistic regression model including the main effects of treatment and center
Statistical Analysis 2: Comparison: Varenicline Tartrate vs Placebo; Week 26; Test type: Superiority or Other; p = 0.0919, Regression, Logistic — p-value obtained from a logistic regression model including the main effects of treatment and center; Missing salivary cotinine was imputed as negative; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.94 to 2.13] — Odds ratio obtained from a logistic regression model including the main effects of treatment and center

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline Tartrate | Placebo
Serious Adverse Events (participants affected / at risk) | 2/213 | 3/218
Other Adverse Events (participants affected / at risk) | 151/213 | 107/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline Tartrate (N=213) | Placebo (N=218)
Cardiac failure (Cardiac disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline Tartrate (N=213) | Placebo (N=218)
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 11 | 5
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 11
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 8 | 8
Flatulence (Gastrointestinal disorders) | 18 | 7
Nausea (Gastrointestinal disorders) | 74 | 14
Vomiting (Gastrointestinal disorders) | 6 | 2
Fatigue (General disorders) | 22 | 15
Irritability (General disorders) | 11 | 9
Pyrexia (General disorders) | 3 | 4
Gastroenteritis (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 7 | 7
Nasopharyngitis (Infections and infestations) | 12 | 8
Pneumonia (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Weight increased (Investigations) | 3 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 1
Disturbance in attention (Nervous system disorders) | 1 | 5
Dizziness (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 22 | 20
Paraesthesia (Nervous system disorders) | 3 | 0
Abnormal dreams (Psychiatric disorders) | 17 | 3
Depressed mood (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 13 | 6
Nightmare (Psychiatric disorders) | 4 | 3
Restlessness (Psychiatric disorders) | 2 | 4
Sleep disorder (Psychiatric disorders) | 22 | 15
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 6
Hypertension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other